CLINICAL TRIAL: NCT04529005
Title: Angiotensin II in the Perioperative Management of Hypotension in Kidney Transplant
Brief Title: Angiotensin II in the Perioperative Management of Hypotension in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Principal Investigator, Scott Benken, Clinical Associate Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0526
Record Dates: First submitted 2020-08-14; First posted 2020-08-27 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Shock, Surgical; Shock; Hypotension and Shock; Kidney Transplant; Complications; Intraoperative Hypotension; Postoperative Hypotension
MeSH Terms: conditions — Shock, Surgical; Shock; Hypotension | interventions — Angiotensin II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Angiotensin II (Giapreza) (Experimental)
  Interventions: Drug: Angiotensin II

INTERVENTIONS:
Drug: Angiotensin II — If intraoperative or postoperative hypotension occurs (e.g. SBP < 120 mmHg) and the attending surgeon and/or attending anesthesiologist deems vasopressor therapy to be necessary, angiotensin II (Giapreza) will be the first vasopressor used for management.

SUMMARY:
The current standard of catecholamine vasopressor management of perioperative hypotension in kidney transplant patients carries significant risks and falls short in many ways. Currently, there is an absence in the scientific literature and research describing the hemodynamic effectiveness and safety of novel pharmacologic agents such as angiotensin II (Giapreza - Ang II) in perioperative kidney transplant patients. Phase 3 registration trials have demonstrated the superior safety and efficacy of Ang II (Giapreza) in distributive shock patients compared to traditional vasopressor agents and the novel mechanism of action may provide additional protection in renal transplant patients. The pilot study entails giving informed and consenting kidney transplant recipients Ang II (Giapreza) as their first vasopressor if the need for vasopressors emerge either intraoperatively or postoperatively in kidney transplant recipients. The primary objective is to evaluate the safety and hemodynamic effects of Ang II (Giapreza) in the renal transplant population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years of age
* Receiving deceased donor kidney transplant
* Pre-transplant Ejection Fraction (within past 18 months) > 50%
* Intraoperative or postoperative distributive shock (according to hospital and study protocol) requiring vasopressor support

Exclusion Criteria:

* Pregnant patients (they would be excluded from receiving a transplant)
* Prisoners
* History of mesenteric ischemia
* History of aortic dissection
* History of abdominal aortic aneurysm
* Allergy to mannitol
* Absolute neutrophil count < 1000 cell/mm3 (within past 18 months)
* Diagnosis of Raynaud's phenomenon, systemic sclerosis or vasospastic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Benken, PharmD, Principal Investigator — Clinical Associate Professor
Locations (1):
- University of Illinois Hospital and Health Sciences System, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aulakh NK, Garg K, Bose A, Aulakh BS, Chahal HS, Aulakh GS. Influence of hemodynamics and intra-operative hydration on biochemical outcome of renal transplant recipients. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):174-9. doi: 10.4103/0970-9185.155144. PMID 25948896
- [Background] Busse LW, Ostermann M. Vasopressor Therapy and Blood Pressure Management in the Setting of Acute Kidney Injury. Semin Nephrol. 2019 Sep;39(5):462-472. doi: 10.1016/j.semnephrol.2019.06.006. PMID 31514910
- [Background] Campos L, Parada B, Furriel F, Castelo D, Moreira P, Mota A. Do intraoperative hemodynamic factors of the recipient influence renal graft function? Transplant Proc. 2012 Jul-Aug;44(6):1800-3. doi: 10.1016/j.transproceed.2012.05.042. PMID 22841277
- [Background] Day KM, Beckman RM, Machan JT, Morrissey PE. Efficacy and safety of phenylephrine in the management of low systolic blood pressure after renal transplantation. J Am Coll Surg. 2014 Jun;218(6):1207-13. doi: 10.1016/j.jamcollsurg.2014.01.058. Epub 2014 Mar 12. PMID 24768292
- [Background] Choi JM, Jo JY, Baik JW, Kim S, Kim CS, Jeong SM. Risk factors and outcomes associated with a higher use of inotropes in kidney transplant recipients. Medicine (Baltimore). 2017 Jan;96(1):e5820. doi: 10.1097/MD.0000000000005820. PMID 28072739
- [Background] Ciapetti M, di Valvasone S, di Filippo A, Cecchi A, Bonizzoli M, Peris A. Low-dose dopamine in kidney transplantation. Transplant Proc. 2009 Dec;41(10):4165-8. doi: 10.1016/j.transproceed.2009.08.058. PMID 20005360
- [Background] Khanna A, English SW, Wang XS, Ham K, Tumlin J, Szerlip H, Busse LW, Altaweel L, Albertson TE, Mackey C, McCurdy MT, Boldt DW, Chock S, Young PJ, Krell K, Wunderink RG, Ostermann M, Murugan R, Gong MN, Panwar R, Hastbacka J, Favory R, Venkatesh B, Thompson BT, Bellomo R, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Deane AM; ATHOS-3 Investigators. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Aug 3;377(5):419-430. doi: 10.1056/NEJMoa1704154. Epub 2017 May 21. PMID 28528561
- [Background] Lankadeva YR, Kosaka J, Evans RG, Bellomo R, May CN. Urinary Oxygenation as a Surrogate Measure of Medullary Oxygenation During Angiotensin II Therapy in Septic Acute Kidney Injury. Crit Care Med. 2018 Jan;46(1):e41-e48. doi: 10.1097/CCM.0000000000002797. PMID 29077618
- [Background] Robert R, Guilhot J, Pinsard M, Longeard PL, Jacob JP, Gissot V, Hauet T, Seguin F. A pair analysis of the delayed graft function in kidney recipient: the critical role of the donor. J Crit Care. 2010 Dec;25(4):582-90. doi: 10.1016/j.jcrc.2010.02.011. Epub 2010 Apr 8. PMID 20381298
- [Background] Toth M, Reti V, Gondos T. Effect of recipients' peri-operative parameters on the outcome of kidney transplantation. Clin Transplant. 1998 Dec;12(6):511-7. PMID 9850443
- [Background] Tumlin JA, Murugan R, Deane AM, Ostermann M, Busse LW, Ham KR, Kashani K, Szerlip HM, Prowle JR, Bihorac A, Finkel KW, Zarbock A, Forni LG, Lynch SJ, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Bellomo R; Angiotensin II for the Treatment of High-Output Shock 3 (ATHOS-3) Investigators. Outcomes in Patients with Vasodilatory Shock and Renal Replacement Therapy Treated with Intravenous Angiotensin II. Crit Care Med. 2018 Jun;46(6):949-957. doi: 10.1097/CCM.0000000000003092. PMID 29509568
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Angiotensin II (Giapreza)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Angiotensin II (Giapreza): The study group received angiotensin II (Giapreza) as the first continuous infusion vasopressor as clinically indicated for either intraoperative or postoperative hypotension not responsive to fluids or push dose vasopressors (intraoperative only).
Arm/Group | Angiotensin II (Giapreza)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6
  Black | 7
  Hispanic | 5
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Duration of ATII Vasopressor Usage in the Intraoperative Setting
Description: Duration of vasopressor usage while in the operating room measured in hours of usage presented as median and IQR.
Time Frame: Duration of usage during the transplant surgery - presented in hours
Population: Started ATII intraoperatively
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Angiotensin II (Giapreza)
Number analyzed (Participants) | 16
hours | 1 [0.5 to 2]

2. Secondary Outcome: Number (and Percentage) of Patients With Arrhythmias
Description: The presence of arrhythmia was confirmed via EKG, flowsheet, or note documentation from the electronic medical record.
Time Frame: From date and time of study drug initiation during or after transplant operation until study drug is discontinued up to a maximum of 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Angiotensin II (Giapreza)
Number analyzed (Participants) | 20
Participants | 1

3. Secondary Outcome: Number (and Percentage) of Patients With Peripheral/Visceral Ischemia
Description: The presence of digital or other peripheral/visceral ischemia was captured from reviewing chart documentation for each patient.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Angiotensin II (Giapreza)
Number analyzed (Participants) | 20
Participants | 0

4. Secondary Outcome: Number (and Percentage) of Patients With Thrombosis
Description: Incidence of venous or arterial thrombosis occurring during the hospitalization for kidney transplant (captured by ultrasound or other diagnostic imaging)
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Angiotensin II (Giapreza)
Number analyzed (Participants) | 20
Participants | 0

5. Secondary Outcome: Number (and Percentage) of Patients With Fungal Infections
Description: The presence of post-operative fungal infections were captured prior to discharge as documented by the clinical care team in the electronic medical record.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Angiotensin II (Giapreza)
Number analyzed (Participants) | 20
Participants | 0

6. Secondary Outcome: Number (and Percentage) of Patients With Hyperglycemia
Description: The presence of hyperglycemia was captured for each patient and was determined by those patients requiring the use of an insulin infusion after their transplant surgery.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Angiotensin II (Giapreza)
Number analyzed (Participants) | 20
Participants | 1

7. Secondary Outcome: Number (and Percentage) of Patients With Delayed Graft Function
Description: The presence of Delayed Graft Function was captured for each patient and defined by the need for renal replacement therapy up to 7 days post-operative.
Time Frame: From post-op to 7 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Angiotensin II (Giapreza)
Number analyzed (Participants) | 20
Participants | 2

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Angiotensin II (Giapreza)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angiotensin II (Giapreza) (N=20)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — defined as platelet count <50,000

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT04529005/Prot_SAP_000.pdf